CLINICAL TRIAL: NCT02279225
Title: RANDOMIZED DOUBLE-BLIND CONTROLLED THE USE OF PHOTOTHERAPY IN FIBROMIÁLGICOS WITH TEMPOROMANDIBULAR JOINT DYSFUNCTION
Brief Title: Protocol Phototherapy Treatment for Fibromyalgia and Temporomandibular Joint Dysfunction
Acronym: FM and DTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Mariana Moreira da Silva, RANDOMIZED DOUBLE-BLIND CONTROLLED THE USE OF PHOTOTHERAPY IN FIBROMIÁLGICOS WITH TEMPOROMANDIBULAR JOINT DYSFUNCTION, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: y4tma2ef
Record Dates: First submitted 2014-10-14; First posted 2014-10-31 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-10

CONDITIONS: Pain; Quality of Life
Keywords: Phototherapy; Laser; Fibromyalgia; DTM/ TMD; Pain
MeSH Terms: conditions — Pain; Fibromyalgia | interventions — Phototherapy; Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (P) (Placebo Comparator): Intervention without radiation
  Interventions: Other: Placebo
- phototherapy (FT) (Experimental): Intervention only with phototherapy radiation
  Interventions: Radiation: Group Phototherapy
- phototherapy+Physical activity (FT+A) (Experimental): Intervention associated
  Interventions: Radiation: Phototherapy + Physical activity
- Physical activity (A) (Experimental): Intervention with physical activity: the gold standard of treatment in fibromyalgia
  Interventions: Other: Physical activity

INTERVENTIONS:
Radiation: Group Phototherapy
  Arms: phototherapy (FT)
Radiation: Phototherapy + Physical activity
  Arms: phototherapy+Physical activity (FT+A)
Other: Physical activity
  Arms: Physical activity (A)
Other: Placebo
  Arms: placebo (P)

SUMMARY:
Temporomandibular joint dysfunction is described as a multifactorial disease and can be directly linked to other diseases, being of structural factors of the Stomatognathic System or not, such as fibromyalgia. Studies show the interconnection of Temporomandibular Dysfunctions with fibromyalgia. Thus, this project aims to evaluate the effect of Phototherapy on fibromiálgicos patients with temporomandibular dysfunction This is a Randomized, Controlled and double-blind, with the intention to treat. In this way the sample of 61 patients with Fibromyalgia, Temporomandibular joint Dysfunction associated with ages between 35 to 58 years, females who are selected after the inclusion/exclusion criteria, will be randomly distributed in homogeneous groups and the placebo group (P), Phototherapy (FT) group, group of physical activity (A) aerobic and aerobic physical activity + Phototherapy Group (FT + A). Will be used as a means of analysis before and after interventions the following parameters: Pain: clinical evaluation, evaluation of pain by Visual analog scale of pain (EVA), McGill Pain Questionnarire and pressure Algometria. Still we will evaluate the dosage of serotonin, indirectly, by saliva. Quality of life: own illness as questionnaires FIQ (Fibromyalgia Impact Questionnaire), Medical Outcomes Study 36-item Short-Form Health Survey SF-36 and also will assess the quality of sleep, with polysomnography. The treatments will total in 10 sessions held twice a week, and the FT and FT + groups to receive Phototherapy enforcement will be used a portable cluster 9 diodes, where will be delivered 39.3 Joules in tender points of fibromyalgia and TMJ, groups and FT + to carry out aerobic activity in 75% of your MHR for 50 min and the P group will receive the application of Phototherapy of 0 Joules (IE, the equipment does not emit any power). Statistical analysis will be compared using the t test intra-group-Student, one-tail and paired and can be used the Kruskal-Wallis test, the statistical analysis of significance 0.05 for both tests.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Fibromyalgia according to the criteria of the American College of Rheumatology;

  * Clinical diagnosis of TMD by the RDC questionnaire (annex I);
  * Cognitive Level enough to understand the procedures and follow the guidelines that will be passed;
  * People who use drugs corresponding to Fibromyalgia (FM), antidepressant;
  * Class I of angle
  * Consent to participate in the study and sign the consent form post information.

Exclusion Criteria:

* With psychiatric disorders;
* Cognitive Changes;
* People who perform some exercise;
* People who carry out orthodontic treatment;
* Systemic diseases;
* Persons under the age of 35 and more than 58 years.

Ages: 35 Years to 58 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 10 sessions, in 5 weeks, 2 times a week
  The time corresponds to assess changes: Assessed on the first day before the start of the first session and the reassessment is made after the last session, after half an hour of intervention. Assessed with questionnaires, and EVA, and algometry.

SECONDARY OUTCOMES:
Quality of sleep | before and after: 10 sessions in 5 weeks, 2 times a week
  The time corresponds to assess changes: Performs initial assessment a week before the first session and the revaluation performs after a week of the last session. evaluation with polysomnography
Quality of life | 10 sessions, in 5 weeks, 2 times a week
  The time corresponds to assess changes: Assessed on the first day before the start of the first session and the reassessment is made after the last session, after half an hour of intervention. Assessed with questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Mariana Moreira Da Silva, São Caetano do Sul, São Paulo, Brazil

REFERENCES:
- [Derived] da Silva MM, Albertini R, Leal-Junior EC, de Tarso Camillo de Carvalho P, Silva JA Jr, Bussadori SK, de Oliveira LV, Casarin CA, Andrade EL, Bocalini DS, Serra AJ. Effects of exercise training and photobiomodulation therapy (EXTRAPHOTO) on pain in women with fibromyalgia and temporomandibular disorder: study protocol for a randomized controlled trial. Trials. 2015 Jun 4;16:252. doi: 10.1186/s13063-015-0765-3. PMID 26040789